CLINICAL TRIAL: NCT04094454
Title: Intrafractional Vaginal Dilation in Anal Cancer Patients Undergoing Pelvic Radiotherapy - Prospective, Randomized, Two-armed Phase-II-study
Brief Title: Intrafractional Vaginal Dilation in Anal Cancer Patients Undergoing Pelvic Radiotherapy
Acronym: DILANA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juergen Debus (Other)
Responsible Party: Sponsor-Investigator, Juergen Debus, Principal Ivestigator, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RADONK-DILANA-2018
Record Dates: First submitted 2019-09-12; First posted 2019-09-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Anal Cancer
Keywords: female patients; quality of life; vaginal dilator; vaginal fibrosis
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tampon with extended vaginal dilatation (Experimental): Patients in arm A will use a special tampon with extended vaginal dilatation during radiotherapy
  Interventions: Device: special tampon with a diameter of 28mm
- Commercially available tampon (Active Comparator): Patients in Arm B will use a normal commercially available tampon (diameter 12-13mm) during radiotherapy
  Interventions: Device: standard tampon with a diameter of 12-13mm

INTERVENTIONS:
Device: special tampon with a diameter of 28mm — patients will use a special tampon with extended vaginal dilatation (diameter 28mm) during radiotherapy
  Arms: Tampon with extended vaginal dilatation
Device: standard tampon with a diameter of 12-13mm — patients in Arm B will use a normal commercially available tampon (diameter 12-13mm) during radiotherapy
  Arms: Commercially available tampon

SUMMARY:
A commercially available vaginal dilator set will be used as measuring device. The grading of vaginal stenosis will be determined as difference of the diameter of vaginal dilator to the baseline. A reduction of the diameter of <20% is defined as vaginal stenosis Grade 1, a reduction of 20-35% as Grade 2, a reduction of >35-49% as Grade 3 and a reduction >/=50% as Grade 4. The investigators hypothesize that the rate of vaginal stenosis Grade 1 or higher 12 months after radiotherapy is lower in the group using extended vaginal dilation during radiotherapy (Arm A). Rates of vaginal stenosis of 50% have been observed in previous patient collectives and the investigators hypothesize that a reduction to 25% is possible in the experimental group.

DETAILED DESCRIPTION:
The study is designed as a prospective, randomized, two-armed, single-center phase-II-trial. 60 patients will be included in the study. Patients fulfilling the inclusion criteria will be randomized into one of the two arms, which differ only in the diameter of a tampon used for vaginal dilatation during treatment. All patients will receive standard (chemo)radiotherapy with a total dose of 45-50,4 Gy (single dose 1,8-2 Gy) to the pelvic and inguinal (if required) lymphatic drainage with a boost to the anal canal up to 54-60 Gy (single doses 1.8-2.2 Gy). The primary objective is the assessment of the incidence and grade of vaginal fibrosis 12 months after (chemo)radiotherapy for anal cancer depending on the extent of intrafractional vaginal dilatation. Secondary endpoints are clinical symptoms and toxicity according to the Common Toxicity Criteria (CTC) version 5.0, assessment of clinical feasibility of daily use of a tampon for vaginal dilatation, assessment of the compliance for the use of a vaginal dilatator and quality of life assessed with the EORTC-QLQ30/-ANL27 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* Histologically confirmed squamous anal cancer
* Indication for definitive or postoperative radiotherapy
* ECOG 0-2
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* patients refusal or incapability of informed consent
* no vaginal dilatation possible prior to radiation treatment start
* prior pelvic irradiation (if direct field border or even overlap of radiation fields assumed)
* participation in another clinical trial which might influence the results of the DILANA trial
* pregnancy/nursing period or inadequate contraception in women with child bearing potential

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
incidence and grade of vaginal fibrosis | Up to 12 months after start of (chemo)radiotherapy
  during and after radiotherapy, clinical symptoms are assessed and graded

SECONDARY OUTCOMES:
clinical symptoms and toxicity according to the CTC AE version 5.0. criteria | weekly during radiotherapy, at each follow-up visit
  during and after radiotherapy, clinical symptoms are assessed and graded according to the CTC AE v5.0 criteria
clinical feasibility of daily use of a special tampon | continously during radiotherapy
  daily assessment of the clinical feasibility of daily use of a special tampon
assessment of the compliance for the use of a vaginal dilatator | continously at every follow-up visit
  patients will be instructed to use a vaginal dilator 3 times a week, at each follow-up visit patients are asked about the frequency of vaginal dilator use
assessment of quality of life | baseline, 6-8 weeks after and 6/12 months after finishing radiotherapy
  EORTC-QLQ30/-ANL27 questionnaires are used to assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Arians, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arians N, Hafner M, Krisam J, Lang K, Wark A, Koerber SA, Hommertgen A, Debus J. Intrafractional vaginal dilation in anal cancer patients undergoing pelvic radiotherapy (DILANA) - a prospective, randomized, 2-armed phase-II-trial. BMC Cancer. 2020 Jan 21;20(1):52. doi: 10.1186/s12885-020-6547-7. PMID 31964381